CLINICAL TRIAL: NCT02048514
Title: The Nellix® EndoVascular Aneurysm Sealing System for the Treatment of Infrarenal Abdominal Aortic Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N09-01
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Aortic Aneurysm, Abdominal; Endovascular Procedures
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nellix Aneurysm Sealing (Experimental): The Nellix® EndoVascular Aneurysm Sealing System
  Interventions: Device: The Nellix® EndoVascular Aneurysm Sealing System

INTERVENTIONS:
Device: The Nellix® EndoVascular Aneurysm Sealing System

SUMMARY:
The purpose of this clinical study is to evaluate the safety and device performance of the Nellix® EndoVascular Aneurysm Sealing System (Nellix System) for the treatment of infrarenal abdominal aortic aneurysms.

DETAILED DESCRIPTION:
This is a multicenter, multi-country prospective, single-arm, non-randomized clinical trial. The comparative control arm is a combination of patient data drawn from the abdominal aortic aneurysms (AAA) open surgical control arms of four commercially approved AAA devices as part of the Society of Vascular Surgeons. Patients enrolled in this study will be pre-screened and have a diagnosis of an infrarenal AAA with or without the need for treatment of iliac artery aneurysm, are candidates for endovascular repair, and meet the eligibility criteria. Patients enrolled in the study will participate in follow-up visits 31 days, 6 months and at 1 year following the index procedure. At the follow-up visits there will be a clinical assessment, blood collection, and abdominal CT imaging of the patient.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Informed consent form understood and signed and patient agrees to all follow-up visits
* Is able and willing to comply with clinical follow-up requirements for one year
* Is able and willing to undergo Contrast-Enhanced Spiral CT scans
* Is a candidate for endovascular repair of an infrarenal aortic aneurysm with or without an iliac aneurysm with at least one of the following;

  1. aneurysm ≥ 4.5 cm in diameter, or
  2. aneurysm is twice the diameter of the normal infrarenal aorta, or
  3. aneurysm is growing at a rate of ≥ 10 % per year
* Non-aneurysmal aortic neck length ≥ 5mm below the most inferior renal artery
* Proximal aortic neck diameter between 16 and 36mm
* Aortic neck angulation to the sac ≤ 60
* Common iliac artery diameter 8 to 35mm bilaterally
* Aneurysm blood lumen diameter ≤ 60mm
* Iliac and femoral arteries suitable for endovascular access with the Nellix System

Exclusion Criteria:

* Life expectancy ≤ 1 year
* Dissecting, ruptured, or leaking aneurysm (blood outside the aorta), has sustained recent trauma, is symptomatic, or is non-degenerative
* Aneurysm is thoraco-abdominal, suprarenal and/or mycotic
* Thoracic aneurysm ≥ 4.5cm in diameter
* AAA requires treatment that would result in bilateral occlusion of the internal iliac arteries
* Presence of mural thrombus > 50% circumferentially in aortic neck
* Iliac aneurysm blood lumen diameter > 35mm
* Active infection, vasculitis, or systemic connective tissue disease (e.g., Rheumatoid arthritis, scleroderma, Marfan's syndrome, Ehlers-Danlos disease) at time of procedure
* History of prior treatment of abdominal aortic or iliac artery aneurysm disease
* Femoral or iliac artery occlusive disease such that device delivery is not possible
* Vascular access for delivery of device requires placement of vascular conduit or is through an established vascular graft
* Receiving dialysis
* History of hypercoagulability
* Allergy to IV contrast
* Serum creatinine level >2.0 mg/dL (or equivalent)
* Patient is pregnant or nursing
* Patient is currently enrolled in an investigational drug or device trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety- Number of Major Adverse Events | 30 day
  The primary safety endpoint is defined as the incidence of Major Adverse Events (MAE) through 30 days after the index procedure.
Device Performance | 30 days
  The primary performance endpoint is technical success defined as successful delivery and deployment of the device and freedom from open surgical conversion at 30 days.

SECONDARY OUTCOMES:
All Cause Mortality | 12 months
  Any death occurring during the study period, regardless of cause

CONTACTS AND LOCATIONS:
Locations (4):
- Centro Medico de Cali, Cali, Colombia
- Paul Stradins University Hospital, Riga, Latvia
- Auckland City Hospital, Auckland, New Zealand
- Instituto de Clinicas Y Urologica Tomanaco, Caracas, Venezuela